CLINICAL TRIAL: NCT04718896
Title: A Multicenter, Open-Label, Randomized Study to Assess the Pharmacokinetics, Safety, and Efficacy of Two Doses of Bimekizumab in Adolescent Study Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Assess the Pharmacokinetics, Safety, and Efficacy of Two Doses of Bimekizumab in Adolescent Study Participants With Moderate to Severe Plaque Psoriasis
Acronym: BE CONNECTED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS0020; 2020-001724-34 (EudraCT Number); 2023-509832-24 (Registry Identifier: EU Clinical Trials); U1111-1303-1875 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: bimekizumab; BKZ; adolescent study participants; psoriasis; PSO
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bimekizumab Dose A (Experimental): Study participants randomized to this arm will receive bimekizumab (BKZ) Dose A at pre-specified time points during the study.
  Interventions: Drug: bimekizumab
- Bimekizumab Dose B (Experimental): Study participants randomized to this arm will receive bimekizumab (BKZ) Dose B at pre-specified time points during the study.
  Interventions: Drug: bimekizumab

INTERVENTIONS:
Drug: bimekizumab — Study participants will receive subcutaneously administered bimekizumab (BKZ) at pre-specified time points during the study.
  Other Names: BKZ; UCB4940

SUMMARY:
The purpose of the study is to assess th pharmacokinetics (PK) of bimekizumab administered subcutaneously (sc) in adolescents with moderate to severe plaque psoriasis (PSO).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥12 to less than 18 years of age at the time of signing the informed consent/assent according to local regulation
* Participant has had a diagnosis of moderate to severe plaque psoriasis (PSO) for at least 3 months prior to the Screening Visit and:

  1. Body surface area (BSA) affected by PSO ≥10%
  2. Investigator's Global Assessment (IGA) score ≥3 (on a scale from 0 to 4)
  3. Psoriasis Area and Severity Index (PASI) score ≥12 OR
  4. PASI score ≥10 plus at least 1 of the following:

  i. Clinically relevant facial involvement ii. Clinically relevant genital involvement iii. Clinically relevant hand and foot involvement
* Participant must be candidate for systemic PSO therapy and/or photo/chemotherapy
* Body weight ≥30 kg and body mass index for age percentile of ≥5 at Baseline
* Male or female A female participant will be eligible to participate if she is not pregnant, not breastfeeding, and a woman of childbearing potential (WOCBP) agrees to follow the contraceptive guidance
* Capable of giving/having parent(s) or legal representative provide signed informed consent/assent (where appropriate)

Exclusion Criteria:

* Participant has a presence of guttate, inverse, pustular, or erythrodermic PSO or other dermatological condition that may impact the clinical assessment of PSO
* Participant has a history of inflammatory bowel disease (IBD) or symptoms suggestive of IBD
* History of active tuberculosis unless successfully treated, latent TB unless prophylactically treated
* Participant has an active infection or history of infections (such as serious infection, chronic infections, opportunistic infections, unusually severe infections)
* Participant has laboratory abnormalities at Screening
* Participant has experienced primary failure to one or more interleukin-17 (IL-17) biologic response modifier OR primary failure to more than 1 biologic response modifier other than an IL-17 biologic response modifier
* Presence of active suicidal ideation, or positive suicide behavior
* Participant has been diagnosed with severe depression in the past 6 months

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of bimekizumab at Week 0 | Baseline (Week 0)
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 0.
Plasma concentration of bimekizumab at Week 1 | Week 1
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 1.
Plasma concentration of bimekizumab at Week 4 | Week 4
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 4.
Plasma concentration of bimekizumab at Week 8 | Week 8
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 8.
Plasma concentration of bimekizumab at Week 12 | Week 12
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 12.
Plasma concentration of bimekizumab at Week 16 | Week 16
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 16.
Plasma concentration of bimekizumab at Week 20 | Week 20
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 20.
Plasma concentration of bimekizumab at Week 36 | Week 36
  Blood samples will be collected at pre-specified time points at Week 36 to determine the bimekizumab plasma concentration, if participant is not eligible for the Open-label Extension (OLE) Period at Week 20 or does not wish to continue into the OLE Period.
Plasma concentration of bimekizumab at Week 40 | Week 40
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 40.
Plasma concentration of bimekizumab at Week 64 | Week 64
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 64.
Plasma concentration of bimekizumab at Week 88 | Week 88
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 88.
Plasma concentration of bimekizumab at Week 112 | Week 112
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 112.
Plasma concentration of bimekizumab at Week 124 | Week 124
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 124.
Plasma concentration of bimekizumab at safety follow up (SFU) | Week 140 (SFU)
  Blood samples will be collected at pre-specified time points to determine the bimekizumab plasma concentration at Week 140 (SFU).

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)]
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks.
Percentage of participants with serious TEAEs | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  An serious adverse event (SAE) must meet 1 or more of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious.
  Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks.
Percentage of participants with TEAEs leading to discontinuation of investigational medicinal product (IMP) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks. This measure considers any TEAE leading to permanent discontinuation of IMP regardless of reason.
Percentage of participants with selected safety topics of interest | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Selected safety topics of interest (including infection [serious, opportunistic, fungal, and tuberculosis (TB)], inflammatory bowel disease [IBD], and injection site reactions) with onset occurring from day of first dose through 20 weeks after final dose of IMP adjusted by duration of participant exposure to IMP.
Change from Baseline in vital signs (systolic and diastolic blood pressure) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Blood pressure will be measured in millimeters of mercury (mmHg).
Change from Baseline in vital signs (heart rate or pulse rate) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Heart rate will be measured in beats per minute (beats/min).
Change from Baseline in vital signs (temperature) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Temperature (oral, axillary, otic or non-contact forehead) will be measured in degrees Celsius (°C).
Change from Baseline in physical examination findings reported as TEAEs with onset occurring from day of first dose through 20 weeks after final dose of IMP | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Clinically significant findings or worsening of previous findings since the physical examination at Baseline will be reported as TEAEs with onset occurring from day of first dose through 20 weeks after final dose of IMP.
Change from Baseline in hematology parameters (platelet count) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Platelets will be measured in number of platelets per liter (10^9/L).
Change from Baseline in hematology parameters (mean corpuscular hemoglobin) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Mean corpuscular hemoglobin (HGB) will be measured in picograms (pg).
Change from Baseline in hematology parameters (mean corpuscular volume) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Mean corpuscular volume will be measured in femtolitres (fL).
Change from Baseline in hematology parameters (erythrocytes) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Erythrocytes will be measured in number of red blood cells per liter (10^12/L).
Change from Baseline in hematology parameters (hemoglobin) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Hemoglobin will be measured in grams per liter (g/L).
Change from Baseline in hematology parameters (hematocrit) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Hematocrit will be measured in volume percentage (%) of red blood cells in blood.
Change from Baseline in clinical chemistry parameters (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase will be measured in units per liter (U/L).
Change from Baseline in hematology parameters (basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Basophils, eosinophils, lymphocytes, monocytes, neutrophils and leukocytes will be measured in number of white blood cells per liter (10^9/L)
Change from Baseline in clinical chemistry parameters (calcium, potassium, sodium, blood urea nitrogen, glucose (nonfasting)) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Calcium, potassium, sodium, blood urea nitrogen, and glucose (non fasting) will be measured in millimoles per liter (mmol/L).
Change from Baseline in clinical chemistry parameters (creatinine, total and direct bilirubin) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Creatinine and bilirubin will be measured in micromols per liter (μmol/L).
Change from Baseline in clinical chemistry parameters (total protein) | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Total protein will be measured in milligrams per liters (mg/L).
Change from Baseline in height | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Growth assessment, as assessed by the change from Baseline in height.
Change from Baseline in weight | From day of first dose (Week 0) through 20 weeks after final dose of IMP (up to Week 140)
  Growth assessment, as assessed by the change from Baseline in weight.
Percentage of participants with Psoriasis Area and Severity Index (PASI) 90 response at Week 16 | Week 16
  The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Percentage of participants with Investigator's Global Assessment (IGA) 0/1 (Clear [0]/Almost Clear [1] with at least 2-category improvement from Baseline) response at Week 16 | Week 16
  The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
  IGA response (Clear or Almost Clear) is defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline.
Percentage of participants with Psoriasis Area and Severity Index (PASI) 75 response at Week 4 | Week 4
  The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Percentage of participants with anti-bimekizumab antibody (AbAb) detection prior to investigational medicinal product (IMP) administration | Baseline (Week 0)
  Anti-bimekizumab antibody (AbAb) detection prior to investigational medicinal product (IMP) administration
Percentage of participants with anti-bimekizumab antibody (AbAb) detection following investigational medicinal product (IMP) administration | From Week 1 through 20 weeks after final dose of IMP (up to Week 140)
  Anti-bimekizumab antibody (AbAb) detection following investigational medicinal product (IMP) administration
Change from Baseline in Children's Dermatology Life Quality Index (CDLQI) response at Week 16 | Week 16, compared to Baseline
  The CDLQI is a questionnaire designed to measure the impact of skin diseases on the lives of children. The questionnaire consists of 10 questions that are based on the experiences of children with skin disease. The instrument asks participants about symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and treatment. The questions relate to the impact of the skin disease on the child over the last week, (ie, over the last 7 days). The CDLQI total score ranges from 0 to 30 with higher scores indicating higher impact of skin disease on quality of life (Qol).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (11):
- United States (2):
  - Ps0020 50344, Indianapolis, Indiana
  - Ps0020 50359, Cypress, Texas
- Canada (2):
  - Ps0020 50354, Calgary
  - Ps0020 50357, St. John's
- Ps0020 40645, Frankfurt, Germany
- Poland (6):
  - Ps0020 40626, Bialystok
  - Ps0020 40625, Lodz
  - Ps0020 40396, Rzeszów
  - Ps0020 40335, Warsaw
  - Ps0020 40333, Wroclaw
  - Ps0020 40334, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org